CLINICAL TRIAL: NCT00363597
Title: Intestinal Permeability and Serum Zonulin Concentration in Children/Adolescents With Functional Dyspepsia
Brief Title: Intestinal Permeability in Children/Adolescents With Functional Dyspepsia
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 0606-104
Record Dates: First submitted 2006-08-11; First posted 2006-08-15 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Functional Dyspepsia
Keywords: dyspepsia; gastrointestinal disease; indigestion
MeSH Terms: conditions — Dyspepsia; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main purpose of this study is to evaluate whether intestinal permeability and/or serum zonulin concentration is increased in children/adolescents with functional dyspepsia (FD). The study will also explore the relationships between intestinal permeability, mucosal inflammation and anxiety in FD patients.

DETAILED DESCRIPTION:
Recurrent abdominal pain is a common complaint among school-age children, being present in up to 15% at any given time. It represents the most common chronic pain entity in pediatric patients. The great majority of these patients will have a functional gastrointestinal disorder (FGID). The most common FGID in these patients is functional dyspepsia (FD), defined as upper abdominal pain or discomfort unrelieved by bowel movement and in the absence of a structural or biochemical explanation for the pain. The etiology of FD is multifactorial, including biological factors, and these factors can be viewed within a biopsychosocial model. Biological factors include inflammation, dysmotility and increased visceral sensitivity. These biological factors are influenced by and are interactive with psychosocial factors such as anxiety, depression and social interaction. This study will evaluate intestinal permeability as a measure of barrier dysfunction and investigate the correlations between increased permeability, mucosal inflammation and anxiety scores to provide further insight into the etiology of FD, thereby assisting in the development and selection of treatment modalities.

ELIGIBILITY:
Inclusion Criteria:

* abdominal pain of at least 8 weeks duration and fulfilling Rome II symptom based criteria for functional dyspepsia (patient group only);
* undergoing endoscopy to evaluate FD following demonstration of a lack of clinical response to standard acid reduction therapy (patient group only); and,
* informed permission/assent

Exclusion Criteria:

* previous abdominal surgery;
* any chronic non-gastrointestinal illness requiring regular medical care (e.g. diabetes mellitus, juvenile rheumatoid arthritis, cystic fibrosis, cancer);
* any history of an adverse reaction to lactulose or mannitol;
* any use of antacids or laxatives within 1 week prior to the study;
* any use of steroids, antihistamines or antihistamine-like drugs within 4 weeks prior to the study;
* any use of aspirin is prohibited within one week prior to the study;
* any use of non-steroidal anti-inflammatory drugs (NSAIDs) other than aspirin is restricted within one week prior to the study or at the discretion of the Study Physician;
* any use of antibiotics including neomycin (Mycifradin) within 4 weeks prior to the study;
* pregnancy;
* any current or chronic history within the previous 6 months of gastrointestinal symptoms including abdominal pain or discomfort, nausea, vomiting, bloating, diarrhea or constipation (healthy control group only); or
* non-English speaking

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with chronic abdominal pain.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2006-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
differential sugar absorption test, serum zonulin | 5 hour urine collection after administration of test article, serum collected during study visit

SECONDARY OUTCOMES:
Behavioral Assessment Scale for Children (BASC) anxiety scores | collected during study visit
T-lymphocyte, eosinophil and mast cell densities on duodenal biopsy samples | collected during biopsy, patient group only

CONTACTS AND LOCATIONS:
Overall Officials: Craig A. Friesen, MD, Principal Investigator — The Children's Mercy Hospital and Clinics
Locations (1):
- The Children's Mercy Hospital and Clinics, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Neilan NA, Garg UC, Schurman JV, Friesen CA. Intestinal permeability in children/adolescents with functional dyspepsia. BMC Res Notes. 2014 May 1;7:275. doi: 10.1186/1756-0500-7-275. PMID 24886078